CLINICAL TRIAL: NCT00204100
Title: The Development of Systems for Paraplegic Cycling: Improving Health After Spinal Cord Injury
Brief Title: Paraplegic Cycling: Improving Health After Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Glasgow (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FEScyclingGlasgow; UK EPSRC: GR/R92462/01
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2006-10-12 (Estimated); Status verified 2005-05

CONDITIONS: Spinal Cord Injury
Keywords: paraplegia; spinal cord injury; functional electrical stimulation; cycling; exercise; cardiopulmonary fitness
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia; Motor Activity

INTERVENTIONS:
Device: Surface Functional Electrical Stimulation

SUMMARY:
Surface electrical stimulation has for many years been widely used to retrain paralysed muscle and achieve the functions of standing and stepping. Recently a number of centres have used electrical stimulation of the leg muscles to achieve cycling. During cycling the quadriceps and hamstring muscles (thigh muscles) (and sometimes also the gluteal (buttocks) muscles) are stimulated to obtain a cycling motion. Stimulation is applied using adhesive electrodes placed on the surface of the skin. This form of exercise is known as FES-cycling (FES = Functional Electrical Stimulation).

We have recently carried out a pilot study which investigated the feasibility of lower-limb cycling using electrical stimulation. Cycling is accomplished using a standard recumbent tricycle, which is adapted for the purpose of FES cycling. Three people with a complete spinal cord lesion at level T7-T10 took part in the pilot study. The subjects are now able to cycle continuously and reliably on a tricycle mounted on a cycle trainer for periods of up to 1 hour. The subjects are also able to cycle outside for distances of up to 3 km.

The purpose of the new study is threefold: (i) We wish to develop the equipment and methods for recreational cycling to the stage of a pre-commercial design specification; (ii) The subjects recruited for the project will carry out a progressive, high-intensity cycle-training programme. In Glasgow, 5 paraplegic subjects shall complete the training programme, which will be based at their homes. This will allow us to fully assess the feasibility of recreational FES-cycling, by measuring the power which can be sustained during long periods of cycling, and to measure the impact of the training regime on their quality of life; (iii) We will determine whether the training regime leads to significant improvements in cardiopulmonary fitness, and therefore lower risk of heart disease, and to reductions in the likelihood of the development of pressure sores and fractures.

We hope that this type of exercise will lead to general improvements in the fitness of people who might use the system in future.

DETAILED DESCRIPTION:
Background:

Spinal cord injury (SCI) prevents normal leg exercise which leads to secondary complications, including cardiopulmonary deconditioning, a high incidence of pressure sores, and bone demineralisation. Wheelchair sports do not raise fitness to the level of sedentary non-injured people but it has been shown that cycling via functional electrical stimulation, "FES-cycling", can. Previous studies have been clinic-based; this limits the exercise time and is inappropriate for widespread use. We propose to show that home-based FES-tricycling can be a recreation, and can also lead to significant health benefits.

We will train subjects at home more intensively than in previous studies, to see whether they can cycle useful distances. The effects of this training will be systematically assessed in a Health Study, which will: (i) regularly monitor cardiopulmonary fitness; (ii) make regular tissue measurements related to pressure sore susceptibility, and (iii) measure the effect on bone density. These health measurements will be made at the collaborating clinical centres, i.e. for Glasgow, this will be at the Queen Elizabeth National Spinal Injuries Unit, Southern General Hospital. We will also document the mobile recumbent tricycle system as a design specification, in preparation for commercialisation.

The project will be based around three centres, in London, Glasgow and Nottwil, and brings together an interdisciplinary team of engineers, exercise scientists, therapists and clinicians.

Aims:

Engineering Development. To develop the equipment and methods for recreational cycling to the stage of a pre-commercial design specification.

Training for Recreation. To carry out a progressive, high-intensity FES cycle-training programme. 15 paraplegic subjects (5 at each centre) shall complete the training programme, which is based at their homes. To assess the feasibility of recreational FES-cycling, by measuring the power which can be sustained during long periods of cycling, and to measure the impact of the training regime on their quality of life.

Health and Fitness Study. To assess whether the training regime leads to significant improvements in cardiopulmonary fitness, and therefore lower risk of heart disease, and to reductions in the likelihood of the development of pressure sores and fractures.

ELIGIBILITY:
Inclusion Criteria:

* Complete spinal cord lesion between T3-T12, of at least 1 year duration. Age between 18-65 years No significant medical or psychiatric complications (assessed by clinician). Sufficient range of motion at the joints (assessed by therapist). No excessive spasticity (assessed by therapist). Bone density in necks of femora and upper tibias > 40 - 60 mg/cm3. Willing to attend the clinic and to exercise at home according to the training programme. Having space at home to set up the tricycle ergometer for frequent use.

Exclusion Criteria:

* Bone density in necks of femora and upper tibias < 40 mg/cm3. Unable to transfer safely between wheelchair and tricycle.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 5
Dates: Start 2003-01; Study Completion 2005-05

PRIMARY OUTCOMES:
changes in cardiopulmonary fitness

SECONDARY OUTCOMES:
changes in:
bone mineral density
muscle bulk
peak muscle force
soft tissue distribution
seating pressure
re-oxygenation after ischaemia

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J Hunt, BSc, PhD, DSc, Principal Investigator — University of Glasgow
Locations (2):
- United Kingdom (2):
  - University of Glasgow, Glasgow, Lanarkshire
  - Queen Elizabeth National Spinal Injuries Unit, Glasgow, Lanarkshire